CLINICAL TRIAL: NCT06636539
Title: Prospective Case Collection Study of Contrast-Enhanced Mammography Imaging Acquired on a New Investigational Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-43
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Breast Screening
Keywords: CEM; Contrast-Enhanced Mammography; Contrast; Diagnostic mammogram; Mammography; Mammogram

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CEM Investigational Exam (Experimental)
  Interventions: Device: CEM Software in New Mammography Device

INTERVENTIONS:
Device: CEM Software in New Mammography Device — All subjects enrolled in the study will undergo a CEM exam.

SUMMARY:
This is a prospective, multi-center image case collection study to acquire de-identified contrast-enhanced breast images on a mammography device to support continuing software technology development. Eligible subjects include women at least 35 years old with a suspicious finding or breast abnormality on a screening or diagnostic mammogram who are indicated for a diagnostic exam or a biopsy procedure.

DETAILED DESCRIPTION:
Contrast-Enhanced Mammography (CEM) is intended to be an extension for diagnostic mammography. It is a technique in which digital 2D mammography is supplemented with the use of intravenous iodinated contrast administration to facilitate cancer detection. The imaging acquired under a contrast agent has preferential uptake in regions of increased vascularity providing complement information for diagnosis. The CEM software application that will be tested is similar to the marketed software I-View™ 2.0 and is intended for use as an adjunct following mammography and/or ultrasound exams as a diagnostic work-up to localize and further characterize a known or suspected lesion.

Thus, to assess the clinical efficacy of the Hologic CEM software I-View in a new mammography device, Sponsor is conducting a prospective case collection study to support the verification and validation of image quality assessments.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity.
* Subject is at least 35 years old
* Subject has a suspicious finding or breast abnormality on a screening or diagnostic mammogram and is indicated for a diagnostic exam or a biopsy procedure.
* Subject is able to read, understand, and sign the study-specific informed consent form (ICF) after the nature of the study has been fully explained to them.

Exclusion Criteria:

* Subject is unable or unwilling to undergo informed consent or subject who requires a Legally Authorized Representative (LAR) for Informed Consent.
* Subject has breast implants, cardiac pacemakers, nipple piercings, or IV ports in the mammography field of view in the breast of interest.
* Subject has had an interventional procedure in the same breast as the suspicious finding within the last six (6) months
* Subject is pregnant or presumed to be pregnant.
* Subject is breastfeeding.
* Subject is actively being treated for cancer of any type with chemotherapy
* Subject is suspected to be at risk of complications from the iodinated contrast agent. These include contra-indications of standard iodinated contrast agents, such as the subject having renal insufficiency) and the subject being on dialysis.
* Subject has had a prior reaction to iodinated contrast; thus, a known allergy to iodinated contrast.
* Subject has had a prior reaction to gadolinium contrast agents; thus, a known allergy to gadolinium contrast.
* Subject who, based on the physician's judgment, may be at increased risk for complications associated with renal function, anticoagulant therapy, or bleeding disorders.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis gender biological women
Enrollment: 75 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects (cases) with lesions | 18 months
  Number of subjects with contrast-enhanced breast images containing lesions as assessed by radiologists' image quality review

CONTACTS AND LOCATIONS:
Overall Officials: Chirag Parghi, MD, Principal Investigator — Solis Mammography
Locations (2):
- United States (2):
  - Solis Mammography Memorial Village, Houston, Texas
  - Washington Radiology Sterling, Sterling, Virginia

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and comply with the IRB. The IRB did not approved the secondary use of IPD at the time the protocol was approved.